CLINICAL TRIAL: NCT00002439
Title: Randomized Phase III Vehicle Controlled Trial of ALRT 1057 Topical Gel in Patients With AIDS-Related Kaposi's Sarcoma
Brief Title: A Study of ALRT 1057 Topical Gel in Patients With AIDS-Related Kaposi's Sarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Clinical Research (Industry)
Collaborators: Ligand Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 272A; L1057T-31; 96ACR-LIG1
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: Sarcoma, Kaposi; HIV Infections
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections | interventions — Alitretinoin

INTERVENTIONS:
Drug: Alitretinoin

SUMMARY:
The purpose of this study is to see if ALRT1057 gel is safe and effective in treating Kaposi's sarcoma (KS) when applied to skin .

DETAILED DESCRIPTION:
This is a Phase 3 double-blind study. KS patients are randomized to 1 of 2 treatment arms. They receive either ALRT1057 gel or placebo for 12 weeks. If progressive disease for KS is noted before Week 12, patients are switched to the other blinded treatment arm. If a response or disease progression that has not persisted for at least 4 weeks as of Week 12 occurs, treatment on the blinded arm is continued for up to 4 additional weeks, or until response of disease progression is confirmed. After that time or after 12 weeks of treatment, open-label ALRT1057 may be received.

ELIGIBILITY:
Information not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

REFERENCES:
- [Background] Walmsley S, Northfelt DW, Melosky B, Conant M, Friedman-Kien AE, Wagner B. Treatment of AIDS-related cutaneous Kaposi's sarcoma with topical alitretinoin (9-cis-retinoic acid) gel. Panretin Gel North American Study Group. J Acquir Immune Defic Syndr. 1999 Nov 1;22(3):235-46. doi: 10.1097/00126334-199911010-00004. PMID 10770343